CLINICAL TRIAL: NCT02459860
Title: Programa Esperanza (Project Hope): A Depression Program for Older Latinos With Chronic Medical Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Maria P. Aranda, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AD-1403-13904
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Depression
Keywords: depression; randomized behavioral trial; aged; Latinos; Spanish-speaking; chronic medical conditions
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem Solving Treatment (Experimental): Problem Solving Treatment Individual, face-to-face PST sessions over a span of 8 weeks and 3 monthly booster sessions. The PST protocol is highly structured, time-limited, and manual-driven; sessions include PST hand outs and homework as well as social and behavioral activation strategies.
  Interventions: Behavioral: Problem Solving Treatment
- Enhanced Usual Care (Active Comparator): Enhanced Usual Care EUC patients will receive psychoeducational materials on depression and depression treatment of older persons. EUC patients will continue to receive the full complement of PACE services (medical, rehabilitation, social) including referrals to specialty mental health services, if indicated.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Problem Solving Treatment — Individual, face-to-face PST sessions over a span of 8 weeks will be held at PACE sites. The first session will last one hour while subsequent sessions will last 45 minutes. After the last PST session, each subject will have 3 monthly booster sessions (about 15 minutes). The PST protocol is intended to be highly structured, time-limited, and manual-driven; sessions include PST hand outs and homework as well as social and behavioral activation strategies, i.e., pleasant activities scheduling. All interventionists will document attendance and provide a post-session fidelity summary. 10% of the individual sessions will be videotaped with patient consent to assess fidelity and training needs.
  Other Names: PST
  Arms: Problem Solving Treatment
Behavioral: Enhanced Usual Care — EUC patients will receive psychoeducational materials on depression and depression treatment of older persons. EUC patients will continue to receive the full complement of PACE services (medical, rehabilitation, social) including referrals to specialty mental health services, if indicated.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to determine whether individually-administered Problem Solving Treatment is effective in managing depressive symptomatology in 250 primarily Spanish-speaking Latino patients ≥55 years of age or older with high medical comorbidity. The aim is to test if Programa Esperanza improves: a) problem solving skills and behavior activation; b) depression-related outcomes; and b) physical functioning compared to enhanced usual care over the course of one year.

DETAILED DESCRIPTION:
The primary aim is to test the comparative effectiveness of Programa Esperanza (Project Hope) a short-term culturally-modified psychosocial intervention for primarily Spanish-speaking Latino patients 55 years of age or older with depression and multiple medical conditions-compared to Enhanced Usual Care (EUC), the alternative choice in real-world care. The study will address the following questions:

Primary Research Question: Among 250 low-income, primarily Spanish-speaking Latinos ≥55 years of age with high medical comorbidity, will Programa Esperanza improve: a) problem solving skills and behavior activation; b) depression-related outcomes; and b) physical functioning compared to EUC over the course of one year?

Exploratory Research Questions:

1. Do moderating conditions exist such that the intervention may be more or less effective for some patient subgroups compared to others?
2. Will qualitative reports from our patient population and provider stakeholders provide key insights related to treatment effectiveness, acceptance and satisfaction, as well as adoption of the intervention within the patient-centered medical home (PCMH) setting?
3. Among patients, interventionists, and organization leaders, are there high feasibility, fidelity, and acceptability of training and deployment of nontraditional interventionists to deliver the psychosocial treatment within the PCMH setting?

Randomized Clinical Trial Design. The study will enroll 250 limited-English-speaking Latinos (55+ years) from the AltaMed Program of All Inclusive Care for the Elderly (PACE), a geriatric patient-centered medical home model in Los Angeles County. Subjects who meet PHQ-9 criteria for depression (i.e., score of 8 or greater) will be randomized to one of two study arms: either individually administered Problem Solving Treatment (PST) sessions (n=125) facilitated by bachelor's-level social workers under the supervision of a licensed clinical social worker; or EUC. Data collected at study enrollment will document past and baseline patient characteristics including baseline depression and depression severity scores. Assessment of depression trial outcomes, i.e., depression symptom level (PHQ-9); depression response and remission rates, and will be taken at 3, 6 and 12 months post randomization.

Study Site. AltaMed is a nonprofit, federally-qualified health center and one of the oldest and largest providers of senior care services for older racial/ethnic minorities in the US for over 30 years. The sample will be recruited from enrollees across 8 licensed PACE treatment sites. PACE is an optional, capitated CMS managed care benefit that provides comprehensive medical and social services to frail people who disproportionately rely on Medicaid/Medicare services. Typical of other PACE programs, AltaMed offers a PCMH comprised of intensive health, therapeutic, and social services for adults at risk of nursing home institutionalization.

Study Subjects/ Selection Criteria/ Recruitment and Enrollment. A total of 250 subjects who meet PHQ-9 criteria for depression (> 8 PHQ-9 score) will be selected for this randomized trial. for detecting major depressive disorder for cut-off scores as low as 8. Potential subjects will be selected from the pool of PACE enrollees and identified by AltaMed staff based on routine PHQ-9 screening conducted face-to-face or by telephone. Those who score positive for depression (> 8 PHQ-9 score) will be recruited and consented to participate in the study by either designated AltaMed staff or study research personnel. Inclusion criteria include: English- or Spanish-speaking Latino age 55 years or older; receiving services from any AltaMed PACE site; positive for depression (> 8 PHQ-9 score). In anticipation of attrition, the investigators will over-recruit subjects at enrollment by 10%.

Procedures. Following screening of PACE enrollees by AltaMed staff, PACE study consenters will apprise potential subjects meeting study criteria of the study protocol and their eligibility and will be responsible for the initial consent procedures. Upon documented written consent, research personnel will conduct a face-to-face structured baseline interview as well as review any questions the participant may have regarding informed consent and the study. Randomization will be conducted at the level of the individual subject. Between 1 to 7 days after the baseline interview, the study program coordinator will contact subjects and apprise them of their treatment status in the study.

Comparators. Problem Solving Treatment. Individual, face-to-face PST sessions (as described above) over a span of 8 weeks will be held at PACE sites. The first session will last one hour while subsequent sessions will last 45 minutes. After the last PST session, each subject will have 3 monthly booster sessions (about 15 minutes). The PST protocol is intended to be highly structured, time-limited, and manual-driven; sessions include PST hand outs and homework as well as social and behavioral activation strategies, i.e., pleasant activities scheduling.

Enhanced Usual Care. EUC patients will receive psychoeducational materials on depression and depression treatment of older persons. The materials are based on our prior work and are available in Spanish and English. EUC patients will continue to receive the full complement of PACE services (medical, rehabilitation, social) including referrals to specialty mental health services, if indicated.

Data Collection. Consented patients will receive a 60 minute face-to-face baseline interview before randomization to be conducted by study personnel. Outcome interviews (60 minutes) will be conducted in-person by independent study interviewers. Data will be based on multiple sources: self-report and clinician-rendered diagnoses, anthropometric measures, medical records and claims data extraction.

Qualitative study design and procedures. In order to address our secondary research questions the investigators will conduct in-depth and focus group interviews with our respective stakeholders.

Patients: During the three post baseline assessment (and after the 3-month quantitative data collection) the investigators will conduct an open-ended component to assess more in-depth explorations of the treatment experience, and longer term issues that may emerge with PST or EUC. This component will be administered based on a guide/questioning route designed to collect in-depth information on the feasibility and acceptability of the intervention based on the subject's own perceptions and reactions to treatment. Dropouts as well as completers will be included. Providers (interventionists, AltaMed managers and executive leadership): The investigators will query providers based on a focus group approach: 2 separate groups of 10 persons each.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking Latino age 55 years or older
* receiving services from any AltaMed PACE site
* positive for depression (> 8 PHQ-9 score)

Exclusion Criteria:

* current drinking problems
* disorders with active mania or psychotic symptoms
* cognitive impairment precluding ability to give informed consent or participating in the intervention
* an active medical condition with life expectancy less than 6 months
* anticipated absences or disenrollment from PACE

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-23 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
PHQ-9 | 3-, 6-, and 12 months
  change from initial screening - depressive symptomatology

SECONDARY OUTCOMES:
SCL-20 | 3-, 6-, and 12 months
  change from baseline - depressive symptomatology
Social Problem-Solving Inventory-Revised | 3-, 6-, and 12 months
  change from baseline - social problem solving skills
PEARLS-Behavioral Activation | 3-, 6-, and 12 months
  change from baseline - behavioral activation
Sheehan Disability Scale | 3-, 6-, and 12 months
  change from baseline - disability level
Performance Oriented Mobility Assessments | 3-, 6-, and 12 months
  change from baseline - physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Maria P Aranda, PhD, Principal Investigator — University of Southern California